CLINICAL TRIAL: NCT07117253
Title: Factors Affecting Outcome of Patients With Interstitial Lung Diseases in Respiratory Intensive Care Unit
Brief Title: Interstitial Lung Diseases in Respiratory ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmine Mamdouh Salah, resident of chest department sohag university, Sohag University
Other Study IDs: Soh-Med-24-10-8MS
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Interstitial Lung Diseases
Keywords: interstitial lung diseases; outcome in icu
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is Prospective observational study to analyze the clinical features, risk factors, outcome,mortality rates in interstitial lung diseases patients who required admission in Respiratory ICU

ELIGIBILITY:
Inclusion Criteria:

* Patients who had diagnosis of interstitial lung diseases required admission in respiratory ICU

Exclusion Criteria:

* Patients with respiratory diseases other than ILD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had diagnosis of interstitial lung diseases required admission in respiratory ICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Complications of disease | 1 month after icu admission
Evaluate Length of respiratory ICU stay | 1 month after icu admission
Assess mortality of patients with interstitial lung diseases in respiratory icu. | 1 month after icu admission

IPD SHARING:
Plan to Share IPD: Undecided